CLINICAL TRIAL: NCT01423968
Title: Impact & Time-Course of Effect of Intravenous Lipopolysaccharide Infusion on Skeletal Muscle Protein Turnover and Insulin Sensitivity in Healthy Human Volunteers
Brief Title: Effect of Lipopolysaccharide on Skeletal Muscle Functions
Acronym: LPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B/12/2010
Record Dates: First submitted 2011-08-11; First posted 2011-08-26 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Sepsis
Keywords: Sepsis; Inflammation; Lipopolysaccharide; Muscle protein turnover; Insulin resistance
MeSH Terms: conditions — Sepsis; Inflammation; Insulin Resistance | interventions — Endotoxins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipopolysaccharide infusion (Experimental): Lipopolysaccharide infusion; dosage 4ng/kg body weight
  Interventions: Biological: Lipopolysaccharide infusion
- saline (Placebo Comparator): 0.9% saline infusion
  Interventions: Other: saline

INTERVENTIONS:
Biological: Lipopolysaccharide infusion — Lipopolysaccharide 4 nanogram/kg body weight
  Other Names: Endotoxin
  Arms: Lipopolysaccharide infusion
Other: saline
  Other Names: 0.9% saline infusion
  Arms: saline

SUMMARY:
The investigators aim to examine how the skeletal muscles of the human volunteers respond to experimental septic conditions to aid understanding of muscle wasting and its biology..

Six healthy men aged 18-30 will be randomly assigned to two metabolic study visits. On the first visit, while resting on a bed, they will have four cannulae inserted including one in the upper thigh, for blood sampling and the infusion of insulin, glucose and normal and tracer amino acids (which allow us to measure muscle protein metabolism). Subjects will receive either injection of purified bacterial product called lipopolysaccharide (LPS) to induce flu-like symptoms or normal saline according to randomization followed by a metabolic test to stimulate muscle synthesis and glucose transport. Three small samples of muscle will be obtained under local anaesthetic from the thigh to measure molecular events in muscle. By performing these measurements, the investigators will determine the consequences of LPS on muscle production and carbohydrate metabolism.

DETAILED DESCRIPTION:
During sepsis, the ability of the body to prevent muscle wasting is impaired resulting in loss of skeletal muscle. In addition, skeletal muscle handling of carbohydrate becomes less efficient. These changes could result in delayed recovery, prolonged rehabilitation and in severe cases mortality of patients. It is still unclear how these changes occur in the human skeletal muscles but animal experiments suggest that protein molecules that are released during sepsis are responsible for these changes. Due to the biological differences between animals and humans in metabolic rate and stability, disease susceptibility and response to infection, simple translation of knowledge from animals to patients could be highly misleading. Therefore, we aim to examine how the skeletal muscles of the human volunteers respond to experimental septic conditions.

Following medical screening, six healthy men aged 18-30 will have two metabolic study visits in a random manner. On the first visit, while resting on a bed, they will have four cannulae inserted including one in the upper thigh, for blood sampling and the infusion of insulin, glucose and normal and tracer amino acids (which allow us to measure muscle protein metabolism). Subjects will receive either injection of purified bacterial product called lipopolysaccharide (LPS) to induce flu-like symptoms or normal saline according to randomization followed by a metabolic test to stimulate muscle synthesis and glucose transport. Three small samples of muscle will be obtained under local anaesthetic from the thigh to measure molecular events in muscle. By performing these measurements, we will determine the consequences of LPS on muscle production and carbohydrate metabolism.

ELIGIBILITY:
Inclusion Criteria:

Male 18-30yrs

Exclusion Criteria:

Clotting disorders Metabolic disease e.g. diabetes, thyroid dysfunction Inflammatory conditions e.g. Crohn's Disease Tobacco smoker Cardiac or Renal pathology Respiratory problems including Asthma Active infectious conditions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Protein Turnover (muscle tracer incorporation) | 4 hr following LPS infusion
  incorporation of 1,2 13C-leucine into muscle tissue

SECONDARY OUTCOMES:
Whole body glucose disposal | 4 h Glucose insulin clamp
  Glucose uptake calculated from glucose infused to maintain euglycemia during a constant insulin infusion.
Expression of genes that regulate muscle protein balance and insulin signalling | 4 h following LPS infusion
  Changes in mRNA levels of several transcripts associated with metabolism or muscle growth in skeletal muscle

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Greenhaff, PhD, Principal Investigator — Professor of Muscle Metabolism, University of Nottingham
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom